CLINICAL TRIAL: NCT05064605
Title: Pharmacological Evaluation of Antifungal Drugs in Respiratory Samples of Patiens With Chronic Pulmonary Aspergillosis
Brief Title: Pharmacological Evaluation of Antifungal in Chronic Pulmonary Aspergillosis
Acronym: EPAR-APC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211257
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Chronic Respiratory Disease; Chronic Pulmonary Aspergillosis
Keywords: Sarcoidosis; Chronic obstructive pulmonary disease; Chronic pulmonary aspergillosis
MeSH Terms: conditions — Sarcoidosis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
At present, pulmonary diffusion and target antifungal concentrations for APC in patients with sarcoidosis or chronic obstructive pulmonary disease (COPD) are unknown.

DETAILED DESCRIPTION:
Knowledge of these elements is however an essential prerequisite for optimizing the dosages in these contexts. The main objective of the study is to quantify the diffusion of antifungals in the lower respiratory tract in patients treated for pulmonary aspergillosis in the context of underlying chronic respiratory disease. Determining this level of diffusion will make it possible to deduce the plasma concentrations to be achieved in patients and to identify the molecules with the best diffusion profile. The concentration of antifungals in the lungs will be measured from 3 types of samples:

* Sputum obtained by expectoration. These samples will make it possible to quantify the diffusion at the level of the upper and lower respiratory tree.
* Bronchial aspirations. These samples will make it possible to quantify the diffusion at the level of the deep respiratory tree.
* Bronchoalveolar lavage fluid, which will quantify the diffusion at the level of the deep respiratory tree and the ELF.

Blood samples will be taken simultaneously so as to determine the percentage of diffusion from the plasma to the lung.

All these samples will be taken as part of the standard care of patients, the lung samples having the main use of mycological monitoring, the blood samples having the main use of pharmacological and serological monitoring. Lung samples will also be taken routinely for pharmacological monitoring, in order to measure antifungal concentrations at the site of infection.

Mycological monitoring will consist of measuring the fungal load in the broncho-respiratory secretions as well as carrying out an antifongigram in the event of isolation of Aspergillus spp.

The possible association between plasma and pulmonary concentrations of antifungals on the one hand, and mycological and clinical markers of treatment efficacy on the other hand, will also be investigated. The mycological markers of efficacy will be the results of mycological monitoring (culture of broncho-respiratory secretions and aspergillus serology). The clinical markers will be the pulmonary imaging results obtained as part of the management of these patients. The identification of such combinations should allow target concentrations of antifungals to be defined and, where appropriate, antifungal dosage recommendations specific to the treatment of PCA in patients with chronic respiratory disease to be defined.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Diagnosis of PCA made according to the criteria of Denning et al. Eur Respir J. 2016
* Previously initiated or newly initiated azole antifungal therapy for chronic lung disease complicated by CPA.
* Informed patients who did not object to the use of their data.

Exclusion Criteria:

* Pregnant woman
* Co-medication affecting the pharmacokinetics of antifungal agents:

Enzyme inducing therapy (rifampin, rifabutin, phenytoin, phenobarbital, efavirenz, nevirapine, etravirine, ritonavir in the case of voriconazole) Drugs that may inhibit the metabolism of antifungal drugs (ritonavir and cobicistat for itraconazole and isavuconazole)

* Patients under guardianship/guardianship
* Patients without social security coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic respiratory diseases such as sarcoidosis or chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Ratio of antifungal concentrations in lung samples/plasma samples depending on the type of lung sample (sputum, bronchial aspiration, bronchoalveolar lavage fluid) | At 12 months
  Ratio of antifungal concentrations in lung samples/plasma samples depending on the type of lung sample

CONTACTS AND LOCATIONS:
Overall Officials: Yurdagül Yuzunhan, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Avicenne, Bobigny, France